CLINICAL TRIAL: NCT00257543
Title: SALT - Alternative Donor Bone Marrow and Cord Blood Transplantation for High Risk Sickle Cell Disease
Brief Title: SALT: Alternative Donor Bone Marrow and Cord Blood Transplantation for High Risk Sickle Cell Disease
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ann E. Haight, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 876-2003
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; bone marrow transplant
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm study (Experimental): this is a single arm study
  Interventions: Procedure: Alternative donor bone marrow and cord blood

INTERVENTIONS:
Procedure: Alternative donor bone marrow and cord blood — bone marrow transplant - alternative donors for bone marrow and cord blood transplants

SUMMARY:
We hope to gain valuable information about the safety, success of engraftment, and rates of complications using alternate donor transplantation for children with severe SCD. Crucial information will be also collected about late effects from alternate donor BMT sickle cell, providing valuable information to clinicians and families making decisions among interventions for children with severe sickle cell disease. If successful, alternate donor transplantation in this setting could pave the way to offering curative treatment to many more patients with severe SCD.

DETAILED DESCRIPTION:
Unfortunately, less than 1/4th of patients with severe SCD will have a matched sibling donor that can serve as a BMT donor. This research protocol proposes to study the safety and usefulness of "alternate donor transplant" (using donors other than matched siblings). We will offer this treatment to children with severe sickle cell disease that do not have a matched sibling BMT donor. Alternative donors can be family members who are slightly less than completely matched, unrelated volunteer donors who are completely matched, and donated banked umbilical cord blood that is completely or nearly completely matched.

Alternative donor transplant has been performed commonly in patients with cancer, and also provides curative therapy for several non-malignant diseases (severe immunodeficiency, marrow failure and metabolic storage diseases). Alternate donor transplants carry higher risks of complications, including graft-versus-host disease, infection, and graft failure. Therefore, we will be selective about which patients are invited to participate, limiting eligibility to those patients that have had a severe SCD related problem (rather than those who are doing well and are likely to have few SCD related problems), but excluding patients who have such severe organ damage that they are more likely to die during transplant, and limiting eligibility to a young age group. A multi-step review algorithm that includes internal, local and external expert review has been constructed to provide a thorough, safe and ethical accrual process. We will treat patients using drugs and methods commonly used in alternate donor transplant for other diseases such as leukemia, and incorporate lessons learned from our previous experience in BMT for sickle cell by modifying supportive care measures. Special attention will be given to evaluation of post-BMT effects in this population, as well as potential reasons for adverse effects (such as graft failure).

We think that Atlanta is a particularly good place to study this kind of transplant for several reasons. One reason is experience: our program has transplanted more children with SCD than any other single institution in North America, with excellent outcomes. Additionally, SCD patients in our area often have been treated on a special red cell transfusion program that limits the number of people donating the blood; we think this is likely to reduce the chance of graft failure.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin SS, hemoglobin SC, or hemoglobin S0 thalassemia
* Donor available: Partially (5/6) HLA-matched relative (PMRD), matched (6/6) unrelated marrow donor or umbilical cord (5/6 or 6/6) of appropriate size (see 6.3.2) , using high-resolution HLA typing. Donor must not be homozygous for HgbS and must meet standard donor eligibility criteria of the Blood and Marrow Transplant Program.
* Severe SCD, defined by one of the following (modified Walters criteria):

oPrevious (6 months prior) central nervous system event lasting longer than 24 hours, plus objective imaging evidence of CNS vasculopathy, with or without residual neurologic findings oFrequent (3 per year for 2 years) painful vaso-occlusive episodes (defined as episode lasting 4 hours and requiring hospitalization or outpatient treatment with parenteral narcotics) oRecurrent (3 in lifetime) acute chest syndrome events which have necessitated exchange transfusion or chronic transfusion therapy. Must have failed a good-faith trial of hydroxyurea (failure defined as a reduction of less than 50% in the incidence of vaso-occlusive events over a period of at least 18 months) or have demonstrated an inability to take the drug due to side effects.

oAny combination of 3 acute chest syndrome episodes and vaso-occlusive pain episodes (defined as above) yearly for 3 years. Must have failed a good-faith trial of hydroxyurea (failure defined as a reduction of less than 50% in the incidence of vaso-occlusive events over a period of at least 18 months) or have demonstrated an inability to take the drug due to side effects.

oStage I or II sickle lung disease oRed-cell alloimmunization (2 antibodies) on chronic transfusion therapy

Exclusion Criteria:

oSuitable HLA-identical relative donor is available oBiopsy proven chronic active hepatitis, portal fibrosis, or cirrhosis, or serologic evidence of active hepatitis.

oSCD chronic lung disease stage III (see Appendix) oSevere renal dysfunction defined as <50% of predicted normal GFR for age. oSevere cardiac dysfunction defined as shortening fraction < 25%. oSevere residual neurologic impairment other than hemiplegia alone, defined as full-scale IQ 70, quadriplegia or paraplegia, inability to ambulate, inability to communicate without assistive device, or any impairment resulting in decline of Lansky performance score to <70%.

oCNS event occurring within 6 months prior to transplant oKarnofsky or Lansky functional performance score < 70% (see Appendix) oConfirmed HIV seropositivity. oPatient with unspecified chronic toxicity serious enough to detrimentally affect the patient's capacity to tolerate bone marrow transplantation.

oPatient or patient's guardian(s) unable to understand the nature and risks inherent in the BMT process.

oHistory of lack of compliance with medical care that would jeopardize transplant course.

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2006-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To determine the frequency of donor engraftment after alternate donor transplantation in children with severe sickle cell disease. | 1 year after completion of study accrual

CONTACTS AND LOCATIONS:
Overall Officials: Ann Haight, M.D., Study Chair — Children's Healthcare of Atlanta/Emory University
Locations (1):
- Children's Healthcare of Altanta, Atlanta, Georgia, United States